CLINICAL TRIAL: NCT00315562
Title: Pilot Study of Early Versus Delayed Carotid Endarterectomy (CEA) for Small to Medium-sized Ischemic Stroke Caused by High-grade Carotid Stenosis
Brief Title: Study of Early Versus Delayed Carotid Endarterectomy (CEA) for Small to Medium-sized Ischemic Stroke Caused by High-grade Carotid Stenosis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCSD IRB #060323
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2007-03

CONDITIONS: Stroke; Carotid Stenosis
Keywords: stroke; carotid stenosis; carotid endarterectomy; timing
MeSH Terms: conditions — Stroke; Carotid Stenosis | interventions — Endarterectomy, Carotid

ARMS (2):
- Early (Experimental): Early
  Interventions: Procedure: carotid endarterectomy
- Delayed (Active Comparator): Delayed
  Interventions: Procedure: carotid endarterectomy

INTERVENTIONS:
Procedure: carotid endarterectomy

SUMMARY:
Pilot study of early versus delayed carotid endarterectomy (CEA) for small to medium-sized ischemic stroke caused by high-grade carotid stenosis.

DETAILED DESCRIPTION:
Pilot study of early versus delayed carotid endarterectomy (CEA) for small to medium-sized ischemic stroke caused by high-grade carotid stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older.
* New small to medium-sized ischemic stroke (defined as less than 1/3 of the MCA territory) in the territory of 70% or greater carotid stenosis.
* Women of child-bearing potential will be included only if there is a negative pregnancy test and they agree to birth control during the treatment period.

Exclusion Criteria:

* Patients judged to be a poor surgical candidate by the treating physicians.
* Unstable neurological status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-04; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
modified Rankin Score | 90 days

SECONDARY OUTCOMES:
stroke incidence | 90 days
transient ischemic attack incidence | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Matt B Jensen, MD, Principal Investigator — UCSD
Locations (1):
- UCSD, San Diego, California, United States